CLINICAL TRIAL: NCT06980350
Title: Proposal of a Novel Model for Identifying Complete Response in dMMR Colon Cancer Following Neoadjuvant Immunotherapy
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Pei-Rong Ding, Director of the Department of Colorectal Surgery, Sun Yat-sen University
Other Study IDs: G2023-176-01
Record Dates: First submitted 2025-05-12; First posted 2025-05-20 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: PD-1 Inhibitors — Patients received at least two doses of anti-PD-1 immunotherapy in a neoadjuvant setting.

SUMMARY:
A novel evaluation model for identifying complete response following neoadjuvant immune checkpoint inhibitor therapy therapy in patients with dMMR colon cancer was developed to validated its efficacy in two independent cohorts, and to assessed its feasibility for W&W strategy.

DETAILED DESCRIPTION:
Immunotherapy shows promise as a curative treatment for patients with non-metastatic dMMR CRC, and offers an option of watch-and-wait (W&W) strategy for those achieving clinical complete response (cCR). A recent study has tested this hypothesis and demonstrated that 100% of patients (n=42) with localized dMMR rectal cancer achieved cCR after 6 months of neoICI treatment. These patients were managed with a W&W strategy, and none experienced tumor recurrence over a median follow-up of 26.3 (range 12.4-50.5) months. This result was echoed by our previous studies, in which patients with dMMR rectal cancer who achieved cCR following neoICI demonstrated promising long-term outcomes.

Organ preservation seems promising not only in patients with dMMR rectal cancer, but also in those with dMMR colon cancer who achieve cCR. In the NEOCAP trail, 20 patients with colon cancer were managed with a W&W strategy, with no tumour regrowth observed over a median follow-up of 11.2 (IQR 5.1-17.7) months. However, the application of organ preservation remains a significant challenge in dMMR colon cancers. This is largely attributed to the fact that tumor responses to neoICI are more prone to be underestimated by radiological assessment. Specifically, patients with pCR were often evaluated as having residual diseases on CT scans. In the PICC trail, 80% (24/30) of patients with partial response (PR) were found to achieve pCR after tumor resection. Similarly, in the NICHE-2 study, only 2 out of 75 patients with pCR had a radiological complete response (CR).5 Hence, a more reliable evaluation model to identify pCR after neoICI in dMMR colon cancer is urgently needed.

In the present study, a novel evaluation model for identifying complete response following neoadjuvant immune checkpoint inhibitor therapy therapy in patients with dMMR colon cancer was developed to validated its efficacy in two independent cohorts, and to assessed its feasibility for W&W strategy.

ELIGIBILITY:
Inclusion Criteria:

1. pathologically confirmed colon adenocarcinoma;
2. immunohistochemistry testing as dMMR tumors;
3. received at least two doses of anti-PD-1 immunotherapy in a neoadjuvant setting.
4. received radical surgery.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with dMMR colon cancer receiving neoICI therapy
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Complete response (CR) | 1 year
  Complete response: Pathological complete response and clinical complete response

CONTACTS AND LOCATIONS:
Overall Officials: Peirong Ding, M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No